CLINICAL TRIAL: NCT02588664
Title: Early Supported Discharge for Improving Functional Outcomes After Stroke
Brief Title: Comprehensive Post-Acute Stroke Services
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Duke University (Other); East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00035998; PCS-1403-14532 (Other: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2015-10-23; First posted 2015-10-28 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2020-12

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: Early Supported Discharge; Transitional Care; Post-acute Stroke Care; Pragmatic Trial; Recovery and Rehabilitation; Secondary Prevention
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participating hospitals randomized to the usual care group will provide their usual, post-acute stroke care to their patients.
- COMPASS Intervention (Active Comparator): Participating hospitals randomized to the intervention will change the structure and process for delivery of post-acute stroke care.
  Interventions: Other: COMPASS Intervention

INTERVENTIONS:
Other: COMPASS Intervention — * A Post-Acute Coordinator (PAC) will visit each patient prior to discharge from the hospital.
  * Patient will receive a follow-up telephone call two days after having been discharged.
  * 7-14 days after discharge, the patient will attend post-acute stroke clinic visit and receive an assessment from an Advanced Practice Provider (APP), a brief patient-reported functional assessment to generate an individualized Care Plan, and referrals from an APP. The patient's primary caregiver will be assessed to ensure caregiver availability and ability to support the patient and the caregiver's ability to cope with the new challenges of caregiving.
  * Patient will receive a call at 30 and 60 days post-discharge for follow-up of functional status, recovery, risk factor management and their access or utilization of recommended services.
  Arms: COMPASS Intervention

SUMMARY:
The purpose of this pragmatic study is to investigate whether implementation of a comprehensive post-acute stroke service model that integrates Early Supported Discharge (ESD) and Transitional Care Management (TCM) for stroke survivors discharged home improves functional outcomes post-stroke, reduces caregiver stress, and reduces readmission rates.

DETAILED DESCRIPTION:
Stroke mortality is 20-40% higher in North Carolina (NC) than in the overall United States. After discharge, stroke patients are at high risk for complications. Although a model of stroke post-care (early supported discharge) exists in Europe and Canada, it has not been adapted for and tested in the US, although patients and stakeholders attest that post-acute care does not meet their needs. Transitional care services from hospital to home are now reimbursed by Centers for Medicaid and Medicare Services (CMS), but only for 30 days after discharge. The study team proposed a pragmatic, cluster randomized trial of 41 NC hospitals to determine the effectiveness of COMprehensive Post-Acute Stroke Services (COMPASS), a patient-centered intervention uniting transitional care management services and elements of early supported discharge in stroke patients discharged directly home.

The study team will build on the successful North Carolina Stroke Care Collaborative (NCSCC) registry, a prospective stroke database in which 51 (of 113) hospitals in NC enroll patients. In preparation for COMPASS, the study team engaged these hospitals via webinars. Over 80% of NCSCC hospitals demonstrated an interest in participation and provided letters of support.

The main question of this pragmatic trial is: Does implementation of COMPASS for all stroke patients discharged directly home improve functional outcomes as measured by the Stroke Impact Scale-16 (SIS-16) at 90 days post-stroke? The primary aim is to: compare the COMPASS model versus usual care on stroke survivors' self-reported functional status at 90 days post-stroke. The secondary aims are to determine if the COMPASS model affects: (1) caregiver strain (Modified Caregiver Strain Index); (2) self-reported general health; (3) disability (Modified Rankin Score); (4) self-reported physical activity; (5) depression (PHQ-2); (6) cognition (MoCA 5-min protocol); (7) medication adherence (Morisky Green Levine Scale-4); (8) self-reported falls; (9) self-reported fatigue (PROMIS Fatigue Instrument); (10) satisfaction with care; (11) secondary prevention - home blood pressure monitoring; (12) self-reported blood pressure; (13-15) all-cause hospital readmissions at 30-days, at 90-days and at 1 year after index discharge; (16-17) mortality at 90-days and at 1 year after index discharge; (18-20) healthcare utilization (emergency department visits, admissions to skilled nursing facilities/inpatient rehabilitation facilities); and (21) use of transitional care management billing codes. This study will also evaluate the effectiveness of the COMPASS Intervention in key patient subgroups based on race, sex, age, diagnosis (stroke versus TIA), stroke severity, and type of health insurance.

English and Spanish-speaking patients ages 18 and older who are admitted to a participating hospital with a diagnosis of ischemic or hemorrhagic stroke or transient ischemic attack and discharged from acute care hospitalization to home will be included (about 6,000 patients/year).

Participating hospitals will be randomized (stratified by stroke volume and primary stroke center status) to receive COMPASS or usual care (control group) in Phase 1. In Phase 2, usual care hospitals will cross over to COMPASS, while the early intervention hospitals sustain the intervention using hospital-based resources.

The trial has three integrated intervention components: (1) COMPASS, which combines transitional care services provided by advanced practice providers (APPs) and early supported discharge services coordinated by the Post-Acute Coordinators (PAC); (2) COMPASS-funded post-acute care coordinators who will engage patient and stakeholder communities to improve post-acute stroke comprehensive stroke services; and (3) development of a stroke metrics scorecard for participating sites. Well-trained APPs and coordinators will have access to online learning and ongoing support/consultation from WFBH personnel and board-certified vascular neurologists.

The study team will assess 90-day and 1-year outcomes. Outcomes at 90-days will be assessed by telephone surveyors blinded to patient's group assignment. Patients will be informed about COMPASS in the hospital and can opt out of 90-day phone follow-up at any time. Those who agree to be surveyed will be asked to provide informed consent at the 90-day phone call to collect outcomes data.

This proposal is led by three highly experienced researchers as co-principal investigators. The team includes expertise in stroke care, large clinical trials, biostatistics, managing clinical registries, survey and acquisition of patient or proxy-reported outcomes, community-based practice improvement, building community coalitions to reduce readmissions, claims analyses, registry management, translating evidence into practice with large multi-site collaboratives, and engaging patients and stakeholders in research. The planning phase of this project has been guided by patients and stakeholders. Each community will form a community resource network to advise and support the implementation of COMPASS, provide feedback to the team, and help create sustainability. If the COMPASS model shows effectiveness, engaged patients and stakeholders will be key partners to disseminate and implement COMPASS throughout the state and beyond.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking stroke patients with diagnosis of ischemic stroke, hemorrhagic stroke or TIA who are discharged home from participating hospitals
* Must be 18 years of age and older at the time of the stroke

Exclusion Criteria:

* Excludes subdural or aneurysmal subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6024 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Duncan, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (40):
- United States (40):
  - CHS Stanly, Albemarle, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - UNC Hospital, Chapel Hill, North Carolina
  - CHS Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - CHS Carolinas Medical Center-Mercy, Charlotte, North Carolina
  - CHS University, Charlotte, North Carolina
  - CHS Northeast, Concord, North Carolina
  - Betsy Johnson Hospital, Dunn, North Carolina
  - Morehead Memorial Hospital, Eden, North Carolina
  - Hugh Chatham Memorial Hospital, Elkin, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Pardee Health, Hendersonville, North Carolina
  - Frye Regional Medical Center, Hickory, North Carolina
  - Novant Health Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Ashe Memorial Hospital, Jefferson, North Carolina
  - Vidant Duplin Hospital, Kenansville, North Carolina
  - CHS Kings Mountain, Kings Mountain, North Carolina
  - Lenoir Memorial Hospital, Kinston, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - WFBH Lexington Medical Center, Lexington, North Carolina
  - CHS Lincoln, Lincolnton, North Carolina
  - Novant Health Matthews Medical Center, Matthews, North Carolina
  - CHS Union, Monroe, North Carolina
  - Carteret County General Hospital, Morehead City, North Carolina
  - CHS Blue Ridge, Morganton, North Carolina
  - Northern Hospital of Surry County, Mount Airy, North Carolina
  - Wilkes Regional Medical Center, North Wilkesboro, North Carolina
  - FirstHealth Moore Regional, Pinehurst, North Carolina
  - Washington County Hospital, Plymouth, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - WakeMed Health and Hospital, Raleigh, North Carolina
  - CHS Cleveland, Shelby, North Carolina
  - Alleghany County Memorial Hospital, Sparta, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Vidant Edgecombe Hospital, Tarboro, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available to researchers through the PCORI-Designated Repository in accordance with their Data Sharing Policy.

REFERENCES:
- [Background] Condon C, Lycan S, Duncan P, Bushnell C. Reducing Readmissions After Stroke With a Structured Nurse Practitioner/Registered Nurse Transitional Stroke Program. Stroke. 2016 Jun;47(6):1599-604. doi: 10.1161/STROKEAHA.115.012524. Epub 2016 Apr 28. PMID 27125528
- [Background] Gesell SB, Klein KP, Halladay J, Bettger JP, Freburger J, Cummings DM, Lutz BJ, Coleman S, Bushnell C, Rosamond W, Duncan PW. Methods guiding stakeholder engagement in planning a pragmatic study on changing stroke systems of care. J Clin Transl Sci. 2017 Apr;1(2):121-128. doi: 10.1017/cts.2016.26. Epub 2017 Feb 27. PMID 28649454
- [Background] Duncan PW, Bushnell CD, Rosamond WD, Jones Berkeley SB, Gesell SB, D'Agostino RB Jr, Ambrosius WT, Barton-Percival B, Bettger JP, Coleman SW, Cummings DM, Freburger JK, Halladay J, Johnson AM, Kucharska-Newton AM, Lundy-Lamm G, Lutz BJ, Mettam LH, Pastva AM, Sissine ME, Vetter B. The Comprehensive Post-Acute Stroke Services (COMPASS) study: design and methods for a cluster-randomized pragmatic trial. BMC Neurol. 2017 Jul 17;17(1):133. doi: 10.1186/s12883-017-0907-1. PMID 28716014
- [Background] Johnson AM, Jones SB, Duncan PW, Bushnell CD, Coleman SW, Mettam LH, Kucharska-Newton AM, Sissine ME, Rosamond WD. Hospital recruitment for a pragmatic cluster-randomized clinical trial: Lessons learned from the COMPASS study. Trials. 2018 Jan 26;19(1):74. doi: 10.1186/s13063-017-2434-1. PMID 29373987
- [Background] Bushnell CD, Duncan PW, Lycan SL, Condon CN, Pastva AM, Lutz BJ, Halladay JR, Cummings DM, Arnan MK, Jones SB, Sissine ME, Coleman SW, Johnson AM, Gesell SB, Mettam LH, Freburger JK, Barton-Percival B, Taylor KM, Prvu-Bettger J, Lundy-Lamm G, Rosamond WD; COMPASS Trial.. A Person-Centered Approach to Poststroke Care: The COMprehensive Post-Acute Stroke Services Model. J Am Geriatr Soc. 2018 May;66(5):1025-1030. doi: 10.1111/jgs.15322. Epub 2018 Mar 23. PMID 29572814
- [Background] Andrews JE, Moore JB, Weinberg RB, Sissine M, Gesell S, Halladay J, Rosamond W, Bushnell C, Jones S, Means P, King NMP, Omoyeni D, Duncan PW; COMPASS investigators and stakeholders. Ensuring respect for persons in COMPASS: a cluster randomised pragmatic clinical trial. J Med Ethics. 2018 Aug;44(8):560-566. doi: 10.1136/medethics-2017-104478. Epub 2018 May 2. PMID 29720489
- [Background] Duncan PW, Abbott RM, Rushing S, Johnson AM, Condon CN, Lycan SL, Lutz BJ, Cummings DM, Pastva AM, D'Agostino RB Jr, Stafford JM, Amoroso RM, Jones SB, Psioda MA, Gesell SB, Rosamond WD, Prvu-Bettger J, Sissine ME, Boynton MD, Bushnell CD; COMPASS Investigative Team. COMPASS-CP: An Electronic Application to Capture Patient-Reported Outcomes to Develop Actionable Stroke and Transient Ischemic Attack Care Plans. Circ Cardiovasc Qual Outcomes. 2018 Aug;11(8):e004444. doi: 10.1161/CIRCOUTCOMES.117.004444. PMID 30354371
- [Background] Bettger JP, Jones SB, Kucharska-Newton AM, Freburger JK, Coleman SW, Mettam LH, Sissine ME, Gesell SB, Bushnell CD, Duncan PW, Rosamond WD. Meeting Medicare requirements for transitional care: Do stroke care and policy align? Neurology. 2019 Feb 26;92(9):427-434. doi: 10.1212/WNL.0000000000006921. Epub 2019 Jan 11. PMID 30635495
- [Background] Halladay J, Bushnell C, Psioda M, Jones S, Lycan S, Condon C, Xenakis J, Prvu-Bettger J; COMPASS Investigative Team. Patient Factors Associated With Attendance at a Comprehensive Postacute Stroke Visit: Insight From the Vanguard Site. Arch Rehabil Res Clin Transl. 2019 Dec 21;2(1):100037. doi: 10.1016/j.arrct.2019.100037. eCollection 2020 Mar. PMID 33543066
- [Background] Gesell SB, Halladay JR, Mettam LH, Sissine ME, Staplefoote-Boynton BL, Duncan PW. Using REDCap to track stakeholder engagement: A time-saving tool for PCORI-funded studies. J Clin Transl Sci. 2020 Feb 6;4(2):108-114. doi: 10.1017/cts.2019.444. eCollection 2020 Apr. PMID 32313700
- [Background] Lutz BJ, Reimold AE, Coleman SW, Guzik AK, Russell LP, Radman MD, Johnson AM, Duncan PW, Bushnell CD, Rosamond WD, Gesell SB. Implementation of a Transitional Care Model for Stroke: Perspectives From Frontline Clinicians, Administrators, and COMPASS-TC Implementation Staff. Gerontologist. 2020 Aug 14;60(6):1071-1084. doi: 10.1093/geront/gnaa029. PMID 32275060
- [Background] Gesell SB, Coleman SW, Mettam LH, Johnson AM, Sissine ME, Duncan PW. How engagement of a diverse set of stakeholders shaped the design, implementation, and dissemination of a multicenter pragmatic trial of stroke transitional care: The COMPASS study. J Clin Transl Sci. 2020 Nov 5;5(1):e60. doi: 10.1017/cts.2020.552. PMID 33948280
- [Background] Pastva AM, Coyle PC, Coleman SW, Radman MD, Taylor KM, Jones SB, Bushnell CD, Rosamond WD, Johnson AM, Duncan PW, Freburger JK; COMPASS Investigative Team. Movement Matters, and So Does Context: Lessons Learned From Multisite Implementation of the Movement Matters Activity Program for Stroke in the Comprehensive Postacute Stroke Services Study. Arch Phys Med Rehabil. 2021 Mar;102(3):532-542. doi: 10.1016/j.apmr.2020.09.386. Epub 2020 Oct 22. PMID 33263286
- [Background] Duncan PW, Bushnell C, Sissine M, Coleman S, Lutz BJ, Johnson AM, Radman M, Pvru Bettger J, Zorowitz RD, Stein J. Comprehensive Stroke Care and Outcomes: Time for a Paradigm Shift. Stroke. 2021 Jan;52(1):385-393. doi: 10.1161/STROKEAHA.120.029678. Epub 2020 Dec 22. PMID 33349012
- [Background] Bayliss WS, Bushnell CD, Halladay JR, Duncan PW, Freburger JK, Kucharska-Newton AM, Trogdon JG. The Cost of Implementing and Sustaining the COMprehensive Post-Acute Stroke Services Model. Med Care. 2021 Feb 1;59(2):163-168. doi: 10.1097/MLR.0000000000001462. PMID 33273292
- [Result] Gesell SB, Bushnell CD, Jones SB, Coleman SW, Levy SM, Xenakis JG, Lutz BJ, Bettger JP, Freburger J, Halladay JR, Johnson AM, Kucharska-Newton AM, Mettam LH, Pastva AM, Psioda MA, Radman MD, Rosamond WD, Sissine ME, Halls J, Duncan PW. Implementation of a billable transitional care model for stroke patients: the COMPASS study. BMC Health Serv Res. 2019 Dec 19;19(1):978. doi: 10.1186/s12913-019-4771-0. PMID 31856808
- [Result] Duncan PW, Bushnell CD, Jones SB, Psioda MA, Gesell SB, D'Agostino RB Jr, Sissine ME, Coleman SW, Johnson AM, Barton-Percival BF, Prvu-Bettger J, Calhoun AG, Cummings DM, Freburger JK, Halladay JR, Kucharska-Newton AM, Lundy-Lamm G, Lutz BJ, Mettam LH, Pastva AM, Xenakis JG, Ambrosius WT, Radman MD, Vetter B, Rosamond WD; COMPASS Site Investigators and Teams.. Randomized Pragmatic Trial of Stroke Transitional Care: The COMPASS Study. Circ Cardiovasc Qual Outcomes. 2020 Jun;13(6):e006285. doi: 10.1161/CIRCOUTCOMES.119.006285. Epub 2020 Jun 1. PMID 32475159
- [Derived] Zhang S, Mormer ER, Johnson AM, Bushnell CD, Duncan PW, Wen F, Pathak S, Pastva AM, Freburger JK, Jones Berkeley SB. The association between neighborhood social vulnerability and community-based rehabilitation after stroke. BMC Health Serv Res. 2025 Jan 10;25(1):55. doi: 10.1186/s12913-024-12142-1. PMID 39794769
- [Derived] Jones Berkeley SB, Johnson AM, Mormer ER, Ressel K, Pastva AM, Wen F, Patterson CG, Duncan PW, Bushnell CD, Zhang S, Freburger JK. Referral to Community-Based Rehabilitation Following Acute Stroke: Findings From the COMPASS Pragmatic Trial. Circ Cardiovasc Qual Outcomes. 2024 Jan;17(1):e010026. doi: 10.1161/CIRCOUTCOMES.123.010026. Epub 2024 Jan 8. PMID 38189125
- [Derived] Kucharska-Newton AM, Halladay JR, Psioda MA, Jones SB, Johnson AM, Coleman SW, Cummings DM, Freburger JK, Daras LC, Rosamond WD, Duncan PW, Bushnell CD. Post-acute Ambulatory Care Service Use Among Patients Discharged Home After Stroke or TIA: The Cluster-randomized COMPASS Study. Med Care. 2023 Mar 1;61(3):137-144. doi: 10.1097/MLR.0000000000001798. Epub 2022 Dec 15. PMID 36729552
- [Derived] Lutz BJ, Kucharska-Newton AM, Jones SB, Psioda MA, Gesell SB, Coleman SW, Johnson AM, Radman MD, Levy S, Bettger JP, Freburger JK, Chou A, Celestino J, Rosamond WD, Bushnell CD, Duncan PW. Familial caregiving following stroke: findings from the comprehensive post-acute stroke services (COMPASS) pragmatic cluster-randomized transitional care study. Top Stroke Rehabil. 2023 Jul;30(5):436-447. doi: 10.1080/10749357.2022.2077520. Epub 2022 May 22. PMID 35603644
- [Derived] Bushnell CD, Kucharska-Newton AM, Jones SB, Psioda MA, Johnson AM, Daras LC, Halladay JR, Prvu Bettger J, Freburger JK, Gesell SB, Coleman SW, Sissine ME, Wen F, Hunt GP, Rosamond WD, Duncan PW. Hospital Readmissions and Mortality Among Fee-for-Service Medicare Patients With Minor Stroke or Transient Ischemic Attack: Findings From the COMPASS Cluster-Randomized Pragmatic Trial. J Am Heart Assoc. 2021 Dec 7;10(23):e023394. doi: 10.1161/JAHA.121.023394. Epub 2021 Nov 3. PMID 34730000
- [Derived] Rosamond WD, Kucharska-Newton AM, Jones SB, Psioda MA, Lutz BJ, Johnson AM, Coleman SW, Schilsky SR, Patel MD, Duncan PW. Emergency department utilization after hospitalization discharge for acute stroke: The COMprehensive Post-Acute Stroke Services (COMPASS) study. Acad Emerg Med. 2022 Mar;29(3):369-371. doi: 10.1111/acem.14401. Epub 2021 Nov 1. No abstract available. PMID 34657341
- Available data/document: Full Data Package — https://www.pcori.org/about-us/governance/policy-data-management-and-data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded subsequent stroke (or TIA) events within the study period (N=142)
Groups:
- COMPASS Intervention: Participating hospitals randomized to the intervention will change the structure and process for delivery of post-acute stroke care.
  COMPASS Intervention: *A Post-Acute Coordinator (PAC) will visit each patient prior to discharge from the hospital.
  * Patient will receive a follow-up telephone call two days after having been discharged.
  * 7-14 days after discharge, the patient will attend post-acute stroke clinic visit and receive an assessment from an Advanced Practice Provider (APP), a brief patient-reported functional assessment to generate an individualized Care Plan, and referrals from an APP. The patient's primary caregiver will be assessed to ensure caregiver availability and ability to support the patient and the caregiver's ability to cope with the new challenges of caregiving.
  * Patient will receive a call at 30 and 60 days post-discharge for follow-up of functional status, recovery, risk factor management and their access or utilization of recommended services.
Period: Overall Study
Arm/Group | Usual Care | COMPASS Intervention
Started | 3193 | 2689
Completed | 1832 | 1644
Not Completed | 1361 | 1045
Not completed — Death | 56 | 55
Not completed — Lost to Follow-up | 1305 | 990

BASELINE CHARACTERISTICS:
Population: Subsequent events (i.e. secondary stroke events) were excluded within the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | COMPASS Intervention | Total
Number analyzed (Participants) | 3193 | 2689 | 5882
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (13.9) | 68.0 (13.8) | 67.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1657 | 1300 | 2957
  Male | 1536 | 1389 | 2925
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 71 | 43 | 114
  Not Hispanic or Latino | 3017 | 2500 | 5517
  Unknown or Not Reported | 105 | 146 | 251
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 20 | 38
  Asian | 18 | 7 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 942 | 489 | 1431
  White | 2122 | 2112 | 4234
  More than one race | 5 | 13 | 18
  Unknown or Not Reported | 86 | 46 | 132
Region of Enrollment [Number; unit: participants]
  United States | 3193 | 2689 | 5882
Stroke Diagnosis [Count of Participants; unit: Participants]
  Ischemic Stroke | 1829 | 1563 | 3392
  Transient Ischemic Attack (TIA) | 1149 | 986 | 2135
  Intracerebral Hemorrhage | 107 | 60 | 167
  Stroke, not otherwise specified | 108 | 80 | 188
NIH Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: units on a scale] — The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The median and interquartile values reflect the mild stroke population.
  units on a scale | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
Health Insurance [Count of Participants; unit: Participants]
  Insured | 2823 | 2440 | 5263
  Uninsured | 293 | 230 | 523
  Missing Insurance Status | 77 | 19 | 96

OUTCOME MEASURES:

1. Primary Outcome: Stroke Impact Scale (SIS-16)
Description: 16-item survey to assess the difficulty level of performing basic physical activities; scores range from 0-100; higher scores correspond to more favorable outcomes
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 3476 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1832 | 1644
score on a scale | 79.9 (21.4) | 80.6 (21.1)

2. Secondary Outcome: Modified Caregiver Strain Index
Description: 13-item survey to measure strain that caregivers may experience; scores range from 0-100; higher scores indicate more caregiver burden
Time Frame: post-stroke day 90
Population: Each enrolled patient was asked to identify a caregiver. A total of 4208 caregivers were identified and asked to complete the Caregiver Questionnaire. A total of 1228 caregivers completed the Caregiver Survey. However, to account for missing data, we utilized inverse probability weight to perform the analysis so the final analysis included was 4208 for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 659 | 569
score on a scale | 21.9 (23.1) | 21.9 (23.5)

3. Secondary Outcome: Self-reported General Health
Description: Self-reported general health is a single question to rate their general health. Responses on a 5-point Likert Scale (Excellent, Very Good, Good, Fair, or Poor) will be analyzed as a continuous variable. Scores range from 95-15 with a higher score indicating better health.
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 3169 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1684 | 1485
score on a scale | 65.4 (28.8) | 66.2 (28.8)

4. Secondary Outcome: Modified Rankin Score
Description: to measure the degree of disability or dependence; scores range from 0-6; higher scores correspond to less favorable outcomes
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 3209 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1680 | 1529
score on a scale | 1 [0 to 3] | 1 [0 to 3]

5. Secondary Outcome: Number of Participants Physically Active and Not Physically Active
Description: Participants are asked whether they walked continuously for at least 10 minutes on any of the last seven days, how many of those days they walked continuously for at least 10 minutes and how many minutes they walked, on average, each day. The physical activity endpoint will be self-reported total number of minutes walked during the past seven days.
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 2968 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1552 | 1416
Participants
  Yes Physically Active (150 min/week of physical activity or more) | 488 | 431
  Not Physically Active (Less than 150 min/week of physical activity) | 1064 | 985

6. Secondary Outcome: Number of Participants With or Without Depression
Description: Based on answers to Patient Health Questionnaire 2-Item (PHQ-2) which is a 2-item questionnaire to determine the frequency of depressed mood; scores range from 0-6; higher scores correspond to less favorable outcomes
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 2,774 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1465 | 1309
Participants
  Not Depressed (or a score of 2 or less on PHQ-2) | 1122 | 1025
  Yes Depressed (or a score of 3 or higher on PHQ-2) | 343 | 284

7. Secondary Outcome: Cognition (MoCA 5-min Protocol)
Description: 4-item questionnaire to determine vascular cognitive impairment; scores range from 0-30; higher scores are more favorable
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 2,728 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1441 | 1287
score on a scale | 24.3 (4.5) | 24.3 (4.7)

8. Secondary Outcome: Medication Adherence (Morisky Green Levine Scale-4)
Description: 4 items with yes/no response options; scores range from 0-4; higher scores correspond to less medication adherence
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 2,730 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1439 | 1291
score on a scale | 0 [0 to 1] | 0 [0 to 1]

9. Secondary Outcome: Number of Participants With or Without Falls
Description: Participants are asked 4 questions to determine whether they have fallen (yes versus no) since hospital discharge, whether or not the fall resulted in a doctor/emergency room visit, whether they have fallen multiple times since discharge, and how many times they have fallen since discharge. Analysis of falls will be based on incidence of any fall since hospital discharge (no falls versus at least one fall).
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 3,055 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1598 | 1457
Participants
  Yes - reported at least 1 fall | 334 | 299
  No - No falls reported | 1264 | 1158

10. Secondary Outcome: Self-reported Fatigue (PROMIS Fatigue Instrument)
Description: 4-question instrument to determine level of fatigue; higher scores correspond to less favorable outcomes; The total raw score is obtained by summing individual question scores and has a range of 4-20. For analysis, raw scores are translated into T-scores which range from 33.7 - 75.8. The T-score rescales the raw score into a standardized score with a mean of 50 and a SD of 10.
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 2,721 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1432 | 1289
score on a scale | 51.5 (10.7) | 51.0 (10.9)

11. Secondary Outcome: Satisfaction With Care
Description: 6 questions to determine satisfaction with care; scores range from 0-100; higher scores correspond to higher satisfaction of care
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 2,929 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1530 | 1399
score on a scale | 6.9 (1.5) | 7.0 (1.4)

12. Secondary Outcome: Number of Participants Who Do or Do Not Monitor Blood Pressure at Home
Description: Participants are asked 2 questions to determine whether they monitor their blood pressure at home (yes or no) and, if they answer in the affirmative, how frequently (daily, weekly, and monthly). Home blood pressure monitoring was analyzed as a dichotomous endpoint (monitoring with any frequency versus no monitoring).
Time Frame: post-stroke day 90
Population: Of the 5,882 that were enrolled in the study, 3,033 provided a response to the survey question. However, we utilized inverse probability weight to perform the analysis in a way to account for missing data. The final analysis included 5,882 for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1586 | 1447
Participants
  Yes - Home BP Monitoring (at least monthly) | 1013 | 1040
  No - Home BP Monitoring (at least monthly) | 573 | 407

13. Secondary Outcome: Self-reported Blood Pressure
Description: 1 question to determine self-reported blood pressure. Self-reported systolic and diastolic BP will each be analyzed as a continuous endpoint. In addition, self-reported systolic and diastolic BP will be used to create a dichotomous hypertension endpoint (systolic BP >= 140 versus systolic BP < 140).
Time Frame: post-stroke day 90
Population: Data was not considered reliable and was therefore not used for analysis. Responses to blood pressure was frequently "120 over 80". This response was so frequent that investigative team did not think the data was a valid measured blood pressure.
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Subjects With Claims-based All-cause Hospital Readmissions
Time Frame: post-stroke day 30
Population: Of the enrolled patients, 2,262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants | 103 | 105

15. Secondary Outcome: Number of Subjects With Claims-based All-cause Hospital Readmissions
Time Frame: post-stroke day 90
Population: Of the enrolled patients, 2,262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants | 222 | 210

16. Secondary Outcome: Number of Subjects With Claims-based All-cause Hospital Readmissions
Time Frame: post-discharge year 1
Population: Of the enrolled patients, 2,262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants | 516 | 485

17. Secondary Outcome: Number of Subjects With All-cause Mortality Using NC State Death Index
Description: Deaths within 90 days of index discharge were ascertained from the North Carolina State Death Index as well as insurance claims beneficiary summary files (i.e. FFS Medicare). A death identified in either database is considered a death.
Time Frame: post-stroke day 90
Population: Mortality by 90-days post-stroke according to the NC State Death Index was collected on all 5,882 enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 3193 | 2689
Participants
  Yes - Did Die | 56 | 55
  No - Did Not Die | 3137 | 2634

18. Secondary Outcome: Number of Subjects With All-cause Mortality Using NC State Death Index & Fee-For-Service (FFS) Medicare
Description: Deaths within 1 year of index discharge were ascertained from the North Carolina State Death Index as well as insurance claims beneficiary summary files (i.e. FFS Medicare). A death identified in either database is considered a death.
Time Frame: post-discharge year 1
Population: Of the enrolled patients, 2262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants
  Yes - Did Die | 105 | 91
  No - Did not Die | 1088 | 978

19. Secondary Outcome: Number of Subjects With Claims-based Emergency Department Visits
Time Frame: post-discharge year 1
Population: Of the enrolled patients, 2262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants | 691 | 626

20. Secondary Outcome: Number of Subjects With Claims-based Admissions to Skilled Nursing Facilities (SNF) and Inpatient Rehabilitation Facilities (IRF)
Time Frame: post-discharge year 1
Population: Of the enrolled patients, 2262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants | 142 | 150

21. Secondary Outcome: Number of Subjects With Claims-based Use of Transitional Care Management Billing Codes
Time Frame: post-discharge day 14
Population: Of the enrolled patients, 2262 were linked to Fee-For-Service (FFS) Medicare claims and included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 1193 | 1069
Participants | 239 | 345

22. Other Pre Specified Outcome: Subgroup Analysis: Race
Description: Analyze the main endpoint of the study in white and non-white individuals
Time Frame: post-stroke day 90
Population: This was a Subgroup Analysis: Race
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

23. Other Pre Specified Outcome: Subgroup Analysis: Sex
Description: Analyze the main endpoint of the study in female and male individuals
Time Frame: measured 90 days post-stroke
Population: Subgroup Analysis: sex
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

24. Other Pre Specified Outcome: Subgroup Analysis: Age
Description: Analyze the main endpoint of the study in <45; 45-<55; 55-<65; 65-<75; >=75 individuals
Time Frame: measured 90 days post-stroke
Population: Subgroup Analysis: Age
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

25. Other Pre Specified Outcome: Subgroup Analysis: Diagnosis (Stroke Versus TIA)
Description: Analyze the main endpoint of the study in stroke versus TIA individuals
Time Frame: measured 90 days post-stroke
Population: Subgroup analysis: diagnosis (stroke versus TIA)
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: Subgroup Analysis: Stroke Severity
Description: Analyze the main endpoint of the study in NIHSS=0, NIHSS=1-4, NIHSS>4 individuals
Time Frame: measured 90 days post-stroke
Population: Subgroup analysis: stroke severity
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

27. Other Pre Specified Outcome: Subgroup Analysis: Type of Health Insurance
Description: Analyze the main endpoint of the study in insured and uninsured individuals
Time Frame: measured 90 days post-stroke
Population: Subgroup analysis: type of health insurance
Arm/Group | Usual Care | COMPASS Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was collected up through day 90 for all subjects and up through year 1 for subjects with Fee-for-Service (FFS) Medicare
Description: Only All-Cause Mortality was collected for the study retrospectively using North Carolina State Death Index. Other adverse Events were not collected as COMPASS was a minimal to no risk study.
Arm/Group | Usual Care | COMPASS Intervention
All-Cause Mortality (participants affected / at risk) | 56/3193 | 55/2689
Serious Adverse Events (participants affected / at risk) | 0/3137 | 0/2689
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Only 58% of intervention hospitals staffed TC clinics continuously. Patient-level barriers were also present and included preference to see primary care providers, affordability, and transportation. Only 35% of patients enrolled through Intervention hospitals received the COMPASS TC Intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Informed Consent Form (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02588664/Prot_ICF_001.pdf
  • Statistical Analysis Plan: Phase 1 (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT02588664/SAP_000.pdf
  • Statistical Analysis Plan: Phase 2 (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT02588664/SAP_002.pdf
  • Statistical Analysis Plan: Claims Data (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02588664/SAP_003.pdf